CLINICAL TRIAL: NCT05568134
Title: Correlations Between CGM and Serum Glucose During OGTT Testing for CFRD
Brief Title: Alternate Measures of Glucose During OGTT Testing for CFRD
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 22-020249
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes
Keywords: continuous glucose monitor; oral glucose tolerance test
MeSH Terms: conditions — Cystic Fibrosis | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- OGTT Cohort: All enrolled participants will complete an OGTT.
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — An oral glucose tolerance test will be completed. A fasting glucose will be measured.
  Participants will drink 1.75 g/kg of dextrose (up to a maximum of 75 grams) within 10 minutes. Glucose values will be measured at 1 hour and 2 hours.

SUMMARY:
Although early detection and treatment of cystic fibrosis-related diabetes (CFRD) can lead to significant clinical improvements and prolong life, rates of screening are poor likely due to the burdensome nature of oral glucose tolerance testing (OGTT). The investigators propose to assess the feasibility and accuracy of two screening tools, continuous glucose monitoring (CGM) and a home OGTT kit (GTT@home). If this pilot study reveals acceptable accuracy of either device, this study will allow for future studies exploring home-based OGTT screening.

DETAILED DESCRIPTION:
The investigators hypothesize that there will be strong agreement between plasma glucose and glucose as measured by either CGM or GTT@home at three different timepoints during an OGTT: fasting, 1-hour, and 2-hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* ≥ 10 years of age
* Fluency in written and spoken English as the GTT@Home is currently only available in English

Exclusion Criteria:

* Hospitalization or treatment with IV antibiotics or supraphysiologic glucocorticoids within 4 weeks
* Major medical or psychiatric disorders other than CF
* Use of medications known to impact the accuracy of the Dexcom G7 (hydroxyurea, >2g acetaminophen per day)
* History of severe adhesive reactions that may lead to an inability to tolerate CGM wear

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 15 subjects with cystic fibrosis (CF) over 10 years of age will be approached to participate.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Agreement between plasma glucose, CGM measured glucose using the Dexcom G7, and GTT@home glucose | Fasting glucose before OGTT
  Differences in fasting glucose will be measured by the difference in mg/dl between plasma glucose, CGM measured glucose, and GTT@home measured glucose.
Agreement between plasma glucose, CGM measured glucose using the Dexcom G7, and GTT@home glucose | 1 hour mark in OGTT
  Differences in the 1 hour glucose during the OGTT will be measured by the difference in mg/dl between plasma glucose, CGM measured glucose, and GTT@home measured glucose.
Agreement between plasma glucose, CGM measured glucose using the Dexcom G7, and GTT@home glucose | 2 hour mark in OGTT
  Differences in the 2 hour glucose during the OGTT will be measured by the difference in mg/dl between plasma glucose, CGM measured glucose, and GTT@home measured glucose.

SECONDARY OUTCOMES:
Agreement between the categorical diagnosis of normal glucose tolerance (NGT), impaired glucose tolerance (IGT), indeterminate glycemia (INDET), and CFRD as defined by plasma glucose, CGM glucose, and GTT@home glucose. | Up to 2 hours
  Categorical diagnosis of glucose tolerance as measured by plasma glucose, CGM measured glucose using the Dexcom G7, and GTT@home glucose.
Difference between plasma glucose and CGM measured glucose after the fasting glucose | Up to 20 minutes after the fasting glucose
  Absolute differences between the glucose measurements will be measured in mg/dL
Difference between plasma glucose and CGM measured glucose after the 1 hour mark during the OGTT. | Up to 20 minutes after the 1 hour mark in the OGTT
  Absolute differences between the glucose measurements will be measured in mg/dL
Difference between plasma glucose and CGM measured glucose after the 2 hour mark during the OGTT. | Up to 20 minutes after the 2 hour mark in the OGTT
  Absolute differences between the glucose measurements will be measured in mg/dL
The ability of untrained participants to successfully complete the GTT@home kit without any guidance from the research team | Up to 2 hours
  Number of steps successfully completed as measured by the GTT@home instruction manual.
Impact of wearing a real-time CGM on participants' awareness of the importance of screening for and diagnosing CFRD. | Within 2 weeks after removal of the CGM
  60 minute semi-structured interviews will be conducted with participants. Transcripts will be analyzed using semantic content analysis
Perceived benefits and burdens of CGM use | Within 2 weeks after removal of the CGM
  Participants will complete a CGM Benefits and Burdens survey, a 16-item measure used to assess perceptions of CGM technology in people with type 1 diabetes. Surveys may be completed on paper or online, as per the participant's preference. The survey is scored on a 5-point scale (agree/disagree scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No